CLINICAL TRIAL: NCT03779490
Title: Transcatheter Repair of Tricuspid Regurgitation With Cardioband TR System Post-Market Clinical Follow-Up Study (TriBAND): A European Prospective, Multicenter Post-market Clinical Follow-up Study to Assess Transcatheter Tricuspid Valve Repair With Edwards Cardioband TR System in Patients With Symptomatic Chronic Functional Tricuspid Regurgitation.
Brief Title: Transcatheter Repair of Tricuspid Regurgitation With Edwards Cardioband TR System Post Market Study (TriBAND)
Acronym: TriBAND
Status: Active, not recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-21
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Tricuspid Regurgitation; Tricuspid Insufficiency
Keywords: Edwards Cardioband TR; Annuloplasty; Tricuspid Repair; Tricuspid Valve
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Repair — Transcatheter Tricuspid Valve Repair with Edwards Cardioband TR

SUMMARY:
The purpose of the study is to assess the safety and the effectiveness of the Cardioband Tricuspid Reconstruction System.

DETAILED DESCRIPTION:
The purpose of the study is to assess the safety and the effectiveness of the Cardioband Tricuspid Reconstruction System. This is a multi-center, prospective, single-arm Post-Market Clinical Follow up Study.

ELIGIBILITY:
* Inclusion Criteria:

  * Eighteen (18) years of age or older
  * Moderate or greater functional Tricuspid Regurgitation (TR)
  * Patient is eligible to receive the Edwards Cardioband TR System per the current approved indications for use.
* Exclusion Criteria:

  * Patients deemed anatomically unsuitable for the device by echocardiography
  * Patients in whom transesophageal echocardiography (TEE) is contraindicated
  * Previous tricuspid valve repair or replacement
  * Severe aortic, mitral and / or pulmonic valve stenosis
  * Severe aortic, mitral and / or pulmonic valve regurgitation
  * Renal Insufficiency requiring dialysis or severe kidney renal disease
  * Life expectancy of less than twelve months
  * Patient is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients with chronic functional tricuspid regurgitation (FTR)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure Success | Hospital discharge, 2-7 days post-procedure
  Reduction in severity of Tricuspid Regurgitation at discharge.

SECONDARY OUTCOMES:
Major Adverse Event Rate | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Rates of major adverse
Procedure Success | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Reduction in severity of Tricuspid Regurgitation (TR) severity
Change in Quality of Life - KCCQ | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Improvement in Quality of Life as assessed by KCCQ.
Change in Quality of Life - EQ-5D-5L | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Improvement in Quality of Life as assessed by EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nickenig, MD, Principal Investigator — Universitätsklinikum Bonn, Germany
Locations (14):
- Germany (12):
  - Ulm University, Ulm, Bavaria
  - Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen, North Rhine-Westphalia
  - Herzzentrum der UniKlinik Köln, Cologne, North Rhine-Westphalia
  - Charité - Universitätsmedizin Campus Mitte, Berlin
  - Berlin Charité-Benjamin Franklin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Herzzentrum Universitätsklinik Dresden, Dresden
  - University Hospital Erlangen, Erlangen
  - Universitätsmedizin Göttingen, Herzzentrum Göttingen, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - UKE Hamburg, Hamburg
  - Katholisches Marienkrankenhaus, Hamburg
- Hospital Universitario Ramón y Cahal, Madrid, Spain
- Universitätsspital Bern (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vernikouskaya I, Bertsche D, Rottbauer W, Rasche V. Deep learning-based framework for motion-compensated image fusion in catheterization procedures. Comput Med Imaging Graph. 2022 Jun;98:102069. doi: 10.1016/j.compmedimag.2022.102069. Epub 2022 May 13. PMID 35576863